CLINICAL TRIAL: NCT04477590
Title: Optimizing Exercise Training Effects on Metabolic Syndrome Factors by Altering the Timing of Medication and Meal Ingestion
Brief Title: Interactions of Medicine and Exercise With Meal Timing
Acronym: MMET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Servicio de Salud de Castilla-La Mancha (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DEP2017-83244-R
Record Dates: First submitted 2020-06-28; First posted 2020-07-20 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Metabolic Syndrome, Protection Against; Exercise Training; Metformin; Statins; Angiotensin-Converting-Enzyme Inhibitor; Fasting, Intermittent; Angiotensin Hypertension
Keywords: Cardiorespiratory fitness; Insulin sensitivity; Dyslipidemia; Hypertension
MeSH Terms: conditions — Metabolic Syndrome; Intermittent Fasting; Insulin Resistance; Dyslipidemias; Hypertension | interventions — Exercise; Dosage Forms; Metformin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Intervention Model Description: Cross-over randomized, pretest-posttest control group experimental design.
Who Masked: Participant, Investigator
Masking Description: Habitual medicine will be embedded in bigger capsules along with a placebo to be able to randomly allocate medicine/placebo. The first meal in the morning will be also masked by either providing a non-caloric or caloric vanilla-flavored beverage resulting in the fed/fasted condition in a blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NO EXERCISE TRAINING (No Intervention): 25-32 individuals with metabolic syndrome that will remain sedentary during the 4 months of treatment taking their habitual medication (i.e., blood pressure, glucose, cholesterol, and triglycerides lowering drugs) and meals at the habitual time (CONTROL GROUP).
- EXERCISE TRAINING FED (Experimental): 2 groups of 25-32 individuals with metabolic syndrome that will exercise-train during 16 weeks after ingesting a liquid test meal (500 calls, 50% fat) 30 min before exercise (EXERCISE TRAINING FED).
  Interventions: Drug: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- EXERCISE TRAINING FASTED (Experimental): 2 groups of 25-32 individuals with metabolic syndrome that will exercise-train during 16 weeks after ingestion of a placebo meal (0 kcals) 30 min before exercise (EXERCISE TRAINING FAST).
  Interventions: Drug: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Drug: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — A group will train 30 min after taking their habitual dose of medicine (MEDICATED train) while another group will train after taking a placebo (NON-MEDICATED train) and will receive their medication after training.
  Other Names: Exercise timing with respect to medication (metformin, statins, ARAII/ACEI)
  Arms: EXERCISE TRAINING FASTED; EXERCISE TRAINING FED

SUMMARY:
To analyze the effects of altering the time of ingestion of participants' habitual medication (i.e., metformin, statins, ARAII/IACE) and meals around the time of exercise training (exercise fasted or fed) on the improvement of metabolic syndrome factors (hypertension, insulin sensitivity, dyslipidemia, and obesity). There will be a preliminary study of the effects of training "time-of-day" on the primary study outcomes.

DETAILED DESCRIPTION:
Objective: The purpose is to study in a group of adults with metabolic syndrome and obesity, the effects of altering timing between exercise training, meals, and their habitual medication on the improvement in the factors that compose the metabolic syndrome (i.e., hypertension, insulin resistance, central obesity, and dyslipidemia). The main objective is to find the most productive combination between exercise training and the timing of their habitual pharmacological treatment, and meal ingestion for lowering those factors.

Methods and design: Cross-over randomized double-blinded, pretest-posttest control group experimental design. The project will be developed in a single center with the collaboration of the regional public health system (SECAM). There will be a preliminary study of the effects of training "time-of-day" on three parallel groups of individuals.

Subjects: Will be referred by their primary care physicians to our study unit or recruited by advertisements in local media.

Up to 180 subjects, all of them with metabolic syndrome will be recruited (>25% women).

Measurements:

Specifically, we will study if the cardiovascular and metabolic adaptations to aerobic training that result in amelioration of metabolic syndrome factors are potentiated by correct timming of training, meals, and medicine around exercise training time.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome patients diagnosed according to The International diabetes federation consensus of 2009 (Alberti, et al., Circulation).

Exclusion Criteria:

* Cardiovascular disease or musculo-skeletal that prevents them from being able to perform intense exercise.

  * Respiratory failure
  * Liver o renal disease
  * Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity assessed using intravenous glucose tolerance test | 12 months
  Curves of insulin-mediated glucose clearance, inhibition of lipolysis, and liver glucose output measured with the use of stable isotope infusion.
Post-prandial lipemia assessed by an oral fat tolerance test | 12 months
  Rates of appearance and clearance of liver VLDL-TG, Apolipoprotein B, and fatty acids using stable isotopes.
Blood pressure assessed by ECG-gated automated sphygmomanometer | 12 months
  Determined immediately after treatments and during the following 24-h using ambulatory blood pressure Holter-type monitors.
Glycemic control assessed by 24-h continuous interstitial glucose monitoring | 36 months
  Determined by a patch glucose sensor paired with a glucose monitor.

SECONDARY OUTCOMES:
Body composition. | 12 months
  Determined by bioelectrical impedance to calculate body fat mass and fat free mass.
Body mass index | 12 months
  Determined by body weight (kg) and height (m) to calculate body mass index (kg/m2)
Maximal oxygen consumption during a graded exercise test to exhaustion, assessed by indirect calorimetry | 12 months
  Calculation of cardiorespitarory fitness
Resting metabolic rate assessed by indirect calorimetry while lying after an overnight fast | 12 months
  Using indirect calorimetry and a ventilated canopy system
Maximal rate of fat oxidation assessed by indirect calorimetry during a submaximal exercise test. | 12 months
  Calculated in grams per min during the incremental cycle ergometer test with the use of indirect calorimetry system
24-hour monitoring of blood concentrations of metformin, statins, and angiotensin blockers assessed using gas chromatography-mass spectrometry. | 36 months
  To study the pharmacokinetics of the habitual medicines used by our subjects during the different experimental conditions
The activity of intramuscular proteins (enzymes) involved in energetics assessed using western blots. | 36 months
  Measured in skeletal muscle obtained by percutaneous muscle biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: RICARDO M Mora-Rodriguez, PhD, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- University of Castilla-La Mancha (Exercise Physiology Lab), Toledo, Spain

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request

REFERENCES:
- [Background] Ortega JF, Hamouti N, Fernandez-Elias VE, de Prada MV, Martinez-Vizcaino V, Mora-Rodriguez R. Metformin does not attenuate the acute insulin-sensitizing effect of a single bout of exercise in individuals with insulin resistance. Acta Diabetol. 2014 Oct;51(5):749-55. doi: 10.1007/s00592-014-0580-4. Epub 2014 Mar 29. PMID 24682492
- [Background] Mora-Rodriguez R, Ortega JF, Guio de Prada V, Fernandez-Elias VE, Hamouti N, Morales-Palomo F, Martinez-Vizcaino V, Nelson RK. Effects of Simultaneous or Sequential Weight Loss Diet and Aerobic Interval Training on Metabolic Syndrome. Int J Sports Med. 2016 Apr;37(4):274-81. doi: 10.1055/s-0035-1564259. Epub 2015 Dec 14. PMID 26667921
- [Background] Alvarez-Jimenez L, Moreno-Cabanas A, Ramirez-Jimenez M, Morales-Palomo F, Ortega JF, Mora-Rodriguez R. Effects of statins and exercise on postprandial lipoproteins in metabolic syndrome vs metabolically healthy individuals. Br J Clin Pharmacol. 2021 Mar;87(3):955-964. doi: 10.1111/bcp.14447. Epub 2020 Jul 12. PMID 32598033
- [Background] Mora-Rodriguez R, Ortega JF, Morales-Palomo F, Ramirez-Jimenez M, Moreno-Cabanas A. Effects of statin therapy and exercise on postprandial triglycerides in overweight individuals with hypercholesterolaemia. Br J Clin Pharmacol. 2020 Jun;86(6):1089-1099. doi: 10.1111/bcp.14217. Epub 2020 Feb 18. PMID 31925809
- [Background] Morales-Palomo F, Ramirez-Jimenez M, Ortega JF, Moreno-Cabanas A, Mora-Rodriguez R. Exercise Training Adaptations in Metabolic Syndrome Individuals on Chronic Statin Treatment. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgz304. doi: 10.1210/clinem/dgz304. PMID 31875915
- [Background] Guio de Prada V, Ortega JF, Morales-Palomo F, Ramirez-Jimenez M, Moreno-Cabanas A, Mora-Rodriguez R. Women with metabolic syndrome show similar health benefits from high-intensity interval training than men. PLoS One. 2019 Dec 10;14(12):e0225893. doi: 10.1371/journal.pone.0225893. eCollection 2019. PMID 31821339
- [Background] Moreno-Cabanas A, Ortega JF, Morales-Palomo F, Ramirez-Jimenez M, Mora-Rodriguez R. Importance of a verification test to accurately assess V̇O2 max in unfit individuals with obesity. Scand J Med Sci Sports. 2020 Mar;30(3):583-590. doi: 10.1111/sms.13602. Epub 2019 Dec 11. PMID 31746500
- [Background] Morales-Palomo F, Ramirez-Jimenez M, Ortega JF, Mora-Rodriguez R. Effectiveness of Aerobic Exercise Programs for Health Promotion in Metabolic Syndrome. Med Sci Sports Exerc. 2019 Sep;51(9):1876-1883. doi: 10.1249/MSS.0000000000001983. PMID 31415443
- [Background] Mora-Rodriguez R, Ortega JF, Ramirez-Jimenez M, Moreno-Cabanas A, Morales-Palomo F. Insulin sensitivity improvement with exercise training is mediated by body weight loss in subjects with metabolic syndrome. Diabetes Metab. 2020 Jun;46(3):210-218. doi: 10.1016/j.diabet.2019.05.004. Epub 2019 May 31. PMID 31158474
- [Background] Mora-Rodriguez R, Ortega JF, Morales-Palomo F, Ramirez-Jimenez M. Weight loss but not gains in cardiorespiratory fitness after exercise-training predicts improved health risk factors in metabolic syndrome. Nutr Metab Cardiovasc Dis. 2018 Dec;28(12):1267-1274. doi: 10.1016/j.numecd.2018.08.004. Epub 2018 Aug 23. PMID 30459053
- [Background] Ramirez-Jimenez M, Morales-Palomo F, Ortega JF, Mora-Rodriguez R. Effects of intense aerobic exercise and/or antihypertensive medication in individuals with metabolic syndrome. Scand J Med Sci Sports. 2018 Sep;28(9):2042-2051. doi: 10.1111/sms.13218. Epub 2018 Jun 4. PMID 29771450